CLINICAL TRIAL: NCT01069172
Title: A Prospective, Randomized Study of Cataract Surgery With the Assistance of the OptiMedica Femtosecond Laser System Compared to Standard Surgical Procedure of Continuous Curvilinear Capsulorhexis and Ultrasonic Phacoemulsification
Brief Title: Study of the Femtosecond Laser System as Compared to Continuous Curvilinear Capsulorhexis for Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OMC-C-2.0
Record Dates: First submitted 2010-02-13; First posted 2010-02-17 (Estimated); Results first posted 2014-09-04 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-08

CONDITIONS: Cataract
Keywords: Cataract; Surgery, cataract extraction; Optical devices, laser
MeSH Terms: conditions — Cataract | interventions — Ultrasonography; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FS Laser Surgery (Experimental): For femtosecond laser-assisted cataract surgery group (FS Laser Surgery), subjects will receive capsulotomy, lens segmentation and, at investigator discretion, lens softening using the femtosecond laser device. If necessary, ultrasound (U/S) phacoemulsification will also be applied to facilitate removal of the crystalline lens during cataract surgery.
  Interventions: Device: FS Laser Surgery
- CCC Surgery (Active Comparator): For the continuous curvilinear capsulorhexis (CCC) group (CCC Surgery), subjects will receive the standard of care for CCC and U/S phacoemulsification surgery to facilitate removal of the crystalline lens during cataract surgery.
  Interventions: Procedure: CCC Surgery

INTERVENTIONS:
Device: FS Laser Surgery — The Catalys System is an ophthalmic surgical laser system intended for use in cataract surgery to perform capsulotomy, lens segmentation, and lens softening, which are all part of cataract surgery when this femtosecond laser is used.
  Other Names: OptiMedica Catalys™ Precision Laser System (Catalys System) = femtosecond laser; Alcon Infiniti System = U/S (ultrasound) phacoemulsification system
  Arms: FS Laser Surgery
Procedure: CCC Surgery — Subjects will receive the standard of care for CCC and U/S cataract surgery to facilitate removal of the crystalline lens. CCC is a procedure that is part of cataract surgery.
  Other Names: Alcon Infiniti System = U/S (ultrasound) phacoemulsification system.
  Arms: CCC Surgery

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the OptiMedica Femtosecond Laser System to perform surgical maneuvers used in the treatment of subjects with cataracts. The safety and efficacy will be compared to the standard surgical procedure of continuous curvilinear capsulorhexis (CCC) and ultrasonic phacoemulsification.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to comply with the treatment/follow-up schedule and requirements
* Able to understand and provide written Informed Consent
* ETDRS (Early Treatment of Diabetic Retinopathy Study) visual acuity equal to or worse than 20/32 (best corrected)
* Age between 50 and 80 years old
* Pupil dilates to at least 7 mm
* Subject able to fixate
* Grade 1-4 nuclear sclerotic cataract (Lens Opacities Classification System - LOCS III)
* Axial length between 22 and 26 mm

Exclusion Criteria:

* Pregnant, intending to become pregnant during course of the study, less than 3 months postpartum or less than 6 weeks after completion of breastfeeding
* Participation in a study of another device or drug within 3 months prior to study enrollment or during this study, and as per the Investigator's careful discretion, as long as not contradictory to any of the above criteria
* Any condition which, in the Investigator's opinion, would make it unsafe (for the subject or for the study personnel) to treat the subject as part of this research study or for which cataract surgery is contraindicated
* Anterior chamber depth (anterior corneal surface to anterior capsule margin) less than 2.5 mm via IOL Master (Zeiss).
* History of prior ocular surgery
* History of ocular trauma
* Co-existing ocular disease affecting vision
* History or current use of alpha-1 antagonist medication (e.g., Flomax)
* Known sensitivity to planned concomitant medications

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan F Batlle, MD, Principal Investigator — Laser Center; William W Culberston, MD, Study Director — Bascom Palmer Eye Institute
Locations (1):
- Laser Center, Santo Domingo, Dominican Republic

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects served as their own control. Subjects were to have FS laser surgery in one eye (FS surgery eyes) and CCC with U/S surgery in their fellow eye (CCC surgery eyes). Assignment to one of the two surgery groups (FS or CCC) was randomized.
Pre-assignment Details: 30 subjects were included in the study, but one subject withdrew prior to surgery on their second eye. Baseline and outcome measure analysis was performed on the 29 subjects with both eyes enrolled. Of these 29 subjects, all had FS laser surgery in one eye (29 FS surgery eyes) and CCC with U/S surgery in their fellow eye (29 CCC surgery eyes).
Groups:
- FS Laser Surgery: For femtosecond laser-assisted cataract surgery (FS Laser Surgery), subjects will receive capsulotomy, lens segmentation and, at investigator discretion, lens softening using the femtosecond laser device.
  FS Laser Surgery: The Catalys System is an ophthalmic surgical laser system intended for use in cataract surgery.
- CCC Surgery: Ultrasound (U/S) cataract surgery and continuous curvilinear capsulorhexis (CCC)
  CCC Surgery: Subjects will receive the standard of care for U/S cataract surgery and CCC to facilitate removal of the crystalline lens.
Period: Overall Study
Arm/Group | FS Laser Surgery | CCC Surgery
Started | 30 (30 eyes) | 30 (30 eyes)
Completed | 29 (29 eyes) | 30 (30 eyes)
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population consists of the 29 subjects that had both eyes enrolled. Of these 29 subjects, all had FS laser surgery in one eye (29 FS surgery eyes) and CCC with U/S surgery in their fellow eye (29 CCC surgery eyes).
Groups:
- FS Laser Surgery and CCC Surgery: Each eye underwent either:
  1. Femtosecond assissisted cataract surgery (FS Laser Surgery), subjects will receive capsulotomy, lens segmentation and, at investigator discretion, lens softening using the femtosecond laser device (the Catalys System is used for FS Laser Surgery and is an ophthalmic surgical laser system intended for use in cataract surgery).
     OR
  2. Ultrasound (U/S) cataract surgery and CCC (continuous curvilinear capsulorhexis), subjects will receive the standard of care for U/S cataract surgery and CCC to facilitate removal of the crystalline lens.
Arm/Group | FS Laser Surgery and CCC Surgery
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.1 (5.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Deviation From Intended Capsulotomy Diameter
Description: Capsulotomy diameter measured during surgery for both the experimental and control groups.
Time Frame: Day of Surgery
Population: 29 subjects had FS laser surgery in one eye (29 FS surgery eyes) and CCC with U/S surgery in their fellow eye (29 CCC surgery eyes). Analysis of capsulotomy size was done by eye group.
Measure: Mean (Standard Deviation); unit: μm
Groups:
- CCC Surgery: Ultrasound (U/S) cataract surgery and continuous curvilinear capsulorhexis (CCC).
  CCC and U/S Surgery: Subjects will receive the standard of care for U/S cataract surgery and CCC to facilitate removal of the crystalline lens.
Arm/Group | FS Laser Surgery | CCC Surgery
Number analyzed (Participants) | 29 | 29
μm | 26.8 (24.6) | 339.1 (248.0)

2. Secondary Outcome: Cumulative Dissipated Energy (CDE)
Description: CDE (the amount of ultrasound energy delivered during phacoemulsification of the crystalline lens) used will be measured during surgery. CDE is a unit used for the Alcon Infinity System (the U/S phacoemulsification used in this study). It is not expressed in standard units such as watts or Joules. CDE, which accounts for the power and time of two ultrasound delivery modes (longitudinal and torsional), is calculated as follows:
  CDE = (Phaco time x average phaco power) + (torsional time x average torsional aptitude x 0.4)
  0.4 is a factor representing the approximate reduction of heat dissipated at the incision as compared to conventional phacoemulsification.
Time Frame: Day of Surgery
Population: 29 subjects had FS laser surgery in one eye (29 FS surgery eyes) and CCC with U/S surgery in their fellow eye (29 CCC surgery eyes). Analysis of CDE was done by eye group.
Measure: Mean (Standard Deviation); unit: CDE
Groups:
- CCC Surgery: Ultrasound (U/S) cataract surgery and continuous curvilinear capsulorhexis (CCC).
  CCC Surgery: Subjects will receive the standard of care for U/S cataract surgery and CCC to facilitate removal of the crystalline lens.
Arm/Group | FS Laser Surgery | CCC Surgery
Number analyzed (Participants) | 29 | 29
CDE | 11.58 (8.35) | 18.54 (12.07)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | FS Laser Surgery | CCC Surgery
Serious Adverse Events (participants affected / at risk) | 2/29 | 1/29
Other Adverse Events (participants affected / at risk) | 0/29 | 6/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FS Laser Surgery (N=29) | CCC Surgery (N=29)
Secondary surgical intervention to reposition lens haptic (Eye disorders) | 1 (1) | 0 (0)
Zonular dehiscence requiring anterior vitrectomy (Eye disorders) | 1 (1) | 0 (0)
Elevated IOP requiring treatment (Eye disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FS Laser Surgery (N=29) | CCC Surgery (N=29)
Elevated intraocular pressure (Eye disorders) | 0 (0) | 6 (6)

LIMITATIONS AND CAVEATS:
This evaluation was performed on a relatively small number of patients; assessment of CDE should be repeated in a larger number of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between the PI and the sponsor (or its agents) that restricts the PI's rights to publish trial results, but does not prohibit publication provided that prior written permission from the sponsor has been granted.